CLINICAL TRIAL: NCT06547879
Title: Effect of an Education Program Based on the Roper, Logan, and Tierney Model of Daily Living Activities Supported With Mindfulness on Self Care, Treatment Adherence, and Healthy Lifestyle Behaviors in Hypertensive Individuals
Brief Title: Effect of a Daily Life Activity-Based Awareness Training Program on Hypertensive Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Hacer Oturmaz, Doctoral Student, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: record 4
Record Dates: First submitted 2024-08-04; First posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Hypertension; Cardiovascular Diseases; Self Efficacy; Treatment Adherence and Compliance; Health Behavior
Keywords: Daily living activities; education; healthy living; hypertension; mindfulness; self-care; treatment adherence
MeSH Terms: conditions — Hypertension; Cardiovascular Diseases; Treatment Adherence and Compliance; Health Behavior

STUDY DESIGN:
Intervention Model Description: The study has a parallel two-group, randomized controlled intervention design.
Who Masked: Participant, Outcomes Assessor
Masking Description: Blinding of Participants:
  Blinding of participants means that the individuals taking part in the study are not aware of which group they have been assigned to, whether it is the intervention group or the control group. This helps to prevent bias in their behavior and responses, as they do not know if they are receiving the actual treatment or a placebo.
  Blinding of Outcome Assessors:
  Blinding of outcome assessors involves keeping the individuals who are measuring and assessing the results of the study unaware of which participants belong to the intervention or control group. This is done to ensure that the data collected and the evaluations made are not influenced by any preconceived notions or expectations about the effectiveness of the intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): One session per week; 20 minutes for the training module and 25 minutes for the awareness practice, a total of 45 minutes each week, for a total of 8 weeks.
  Interventions: Behavioral: Hypertension Self Management Program
- Control group (No Intervention): Usual care.

INTERVENTIONS:
Behavioral: Hypertension Self Management Program — The HT self-management training program was continued in the form of one session per week, a total of 8 modules, for 8 weeks, with different module content each week. After these eight-week training and awareness sessions were completed, the implementation of the study was terminated (week 8), no additional intervention was given to the intervention group, and the evaluations at the 8th week (end of intervention-T1) and the 12th week (follow-up-T2) were carried out by the researcher during the routine checks of the participants at the outpatient clinic. It was carried out face to face.
  Arms: Intervention group

SUMMARY:
This randomized controlled study evaluated an education program based on the Roper, Logan, and Tierney model of daily living activities, supported by mindfulness, for hypertensive individuals. The intervention group received eight weeks of online sessions, while the control group received routine care. Results showed significant improvements in systolic and diastolic blood pressure, self-care, treatment adherence, and healthy lifestyle behaviors in the intervention group compared to controls (p<0.05). Findings suggest that mindfulness-supported education enhances hypertension management. Further studies with larger samples and long-term follow-up are recommended.

DETAILED DESCRIPTION:
Considering that theory-based educational practices alone are not sufficient in the management of HT and that a multifaceted perspective must be developed, in addition to the education based on the ADL nursing model, the conscious awareness approach, which is effective in stress management with its easy integration into daily life, has also been included in this program. In this way, individuals can gain experience and reach self-awareness as a result of theory and skill-based training and feel more motivated to adopt healthy lifestyle behaviors. Multicomponent interventions offer a more comprehensive approach by combining a variety of methods, such as mindfulness, exercise, and dietary changes, as well as educational programs. Such integrated interventions can positively impact both individuals' knowledge and lifestyle habits, providing more effective results in the management of HT and contributing to long-term health improvements.

In this context, this study aimed to evaluate the effect of the training program, structured according to Roper, Logan and Tierney's ADL nursing model and supported by awareness, on self-care, treatment compliance and healthy lifestyle behaviors in individuals with HT. This research is the first randomized controlled study in which the effects of a training program that is suitable for our country's patient profile for HT self-management, shaped according to multidimensional and up-to-date guidelines, that can encourage participants to change behavior, are tested. It has the potential to provide unique contributions to the field with its potential to create infrastructure.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 65
* Literate (able to read and write)
* Followed up for at least 6 months with a diagnosis of stage 1 primary hypertension (HT)
* Taking at least one antihypertensive medication
* No changes in antihypertensive medication in the past month
* Able to use a smartphone and WhatsApp® application
* Having internet access and willing to participate in online sessions

Exclusion Criteria:

* Those with hearing and vision problems
* Those with cognitive impairment
* Having a psychiatric diagnosis such as major depression
* Having a history of major heart surgery in the last 6 months
* Those with severe symptom burden due to advanced COPD, heart failure, asthma, cancer
* Individuals who used another mind-body-based approach (yoga, meditation, relaxation exercise, etc.) during the research were not included in the sample.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2023-03-15 (Actual); Primary Completion 2023-05-15 (Actual); Study Completion 2024-07-05 (Actual)

PRIMARY OUTCOMES:
Hypertension Self-Care Profile | At week 0, week 8 and week 12
  The Hypertension Self-Care Profile Scale has three subscales: behavior, motivation and self-efficacy. In this scale, each sub-dimension is evaluated separately and a total of minimum 20 and maximum 80 points can be obtained from the scale. Higher scores indicate better self-care.
Hill-Bone Hypertension Treatment Compliance Scale | At week 0, week 8 and week 12
  The scale consists of three sub-dimensions (interview, medical and nutrition) and a total of 14 questions. The total score that can be obtained from the scale varies between 14 and 56; A score of 14 indicates full compliance, while higher scores indicate treatment non-compliance.
Healthy Lifestyle Behaviors Scale II | At week 0, week 8 and week 12
  It aims to evaluate individuals' behaviors towards healthy lifestyles. There are 52 items in total in the scale, and all of the items consist of positive expressions. The minimum score that can be obtained from the scale is 52 and the maximum score is 208.
Conscious awareness | At week 0, week 8 and week 12
  It evaluates individual differences in individuals' states of consciousness and measures their tendency to be aware of and pay attention to momentary experiences in daily life. The total score that can be obtained varies between 15 and 90. A high score indicates a high level of conscious awareness.

SECONDARY OUTCOMES:
Systolic and diastolic blood pressure | At week 0, week 8 and week 12
  Blood pressure measurement by the researcher with a digital device.
Metabolic Control Variables | At week 0 and week 8
  A total of 15 items regarding fasting blood sugar, HbA1c, urea, creatinine, uric acid, glomerular filtration rate, serum sodium and potassium values, lipid panel, hemogram, height, weight and BMI values.
Hypertension Information Assessment | At week 0 and week 8
  Individuals' HT knowledge status before and after the intervention was evaluated and the data were classified as "correct" and "incorrect" and calculated as number-percentage.

CONTACTS AND LOCATIONS:
Overall Officials: Hacer Eroğlu, Principal Investigator — haceroturmaz@hacettepe.edu.tr
Locations (1):
- Ornek Mahallesi, 2061. Caddesi 4/1 Blok No:37, Altındağ, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Researchers interested in accessing the IPD should contact the study's principal investigator via email at [email address]. Requests will be reviewed and responded to within four weeks.